CLINICAL TRIAL: NCT01412905
Title: Telemedicine Retinal Screening Utilizing a Mobile Medical Unit With a Trained Technician Accurately Detects Disease in High Risk Ethnically Diverse Populations: Results of a Project Dulce™ Retinal Screening Study
Brief Title: Telemedicine Retinal Screening Utilizing a Mobile Medical Unit
Status: Completed | Type: Observational
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: Fonseca Family Foundation (Unknown); Blue Shield Foundation (Unknown); NCRR 1U54RR025204-01-01 (Unknown)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corp VP, Scripps Whittier Diabetes Institute
Other Study IDs: SWDI-Retinal
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Diabetes; Retinopathy
Keywords: screening; diabetic retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Retinal Diseases; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Objective: To test the accuracy of a referral system for diabetic eye disease conducted by a trained screener using a digital camera, a mobile medical unit and a centralized image-storing software in underserved, ethnically diverse neighborhoods in San Diego.

Methods and Research Design: Retinal screening exams were offered at 8 community health centers for 1229 individuals, ages 16-80 years with diabetes throughout San Diego County over 18 months. Images were captured with a special digital camera, securely transferred to a software system and read independently by a trained technician and retinal specialist. An analysis was conducted to evaluate who had severe eye disease and how accurate the reading of the technician were compared to the expert ophthalmologist readings.

The investigators would like to demonstrate that telemedicine retinal screening utilizing a mobile medical unit with a trained technician in high-risk, ethnically diverse populations can accurately detect positive and negative disease. This may be a model to increase access to retinal examination in order to meet current guidelines and can allow more efficient use of the retinal specialist to evaluate and treat disease leading to a more cost efficient method of care.

DETAILED DESCRIPTION:
Objective: To test the validity and accuracy of a grading and referral system for diabetic retinopathy conducted by a trained screener using a digital camera, a mobile medical unit and a centralized image-storing software in underserved, ethnically diverse neighborhood community health centers Methods and Research Design: Retinal screening exams using telemedicine technology were offered at 8 community health centers for 1229 individuals, ages 16-80 years with diabetes throughout San Diego County over 18 months. Images were electronically captured, transferred to EyePACs1 image software and read independently by a trained technician and retinal specialist. Statistical analysis was conducted to evaluate prevalence of disease and accuracy and validity of readings. Snellen eye test and glaucoma testing using tonometry will also be conducted.

Results: Will evaluate demographics that include age, gender, ethnicity, duration of diabetes, type of diabetes and need for dilation. Severity of disease will be captured. Statistical analysis will be conducted for technician accuracy of grading the readings.

Conclusions: To demonstrate that telemedicine retinal screening utilizing a mobile medical unit with a trained technician in high-risk, ethnically diverse populations can accurately detect positive and negative screens. This may be a model to increase access to retinal examination in order to meet ADA and HEDIS guidelines and can allow more efficient use of the retinal specialist to evaluate and treat disease leading to a more cost efficient method of care.

ELIGIBILITY:
Inclusion Criteria:

* age 16-80 years;
* diagnoses of type 1 or 2 diabetes;
* enrolled in one of the participating clinics or has a personal primary care provider;
* no or minimal insurance and is a San Diego County resident.

Exclusion criteria:

* high intra-ocular pressure > 21 mmHg and < 4 mm of pupil dilation
* known allergy to latex .

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and Women, ages 16-80 with type 1 and type 2 diabetes mellitus identified from 8 community health centers in San Diego County.
Sampling Method: Non-Probability Sample
Enrollment: 1229 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute
Locations (1):
- Scripps Whittier Diabetes Institute, La Jolla, California, United States